CLINICAL TRIAL: NCT03482492
Title: Comparison of Tramadol vs. Tramadol With Paracetamol for Efficacy of Postoperative Pain Management in Lumbar Discectomy: A Randomised Controlled Trial
Brief Title: Tramadol vs.Tramadol With Paracetamol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University Hospital (Other)
Responsible Party: Principal Investigator, Neslihan Uztüre, Principal Investigator, Yeditepe University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 11.03.2014-397
Record Dates: First submitted 2018-03-20; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Lumbar Disc Herniation
Keywords: Acetaminophen; Tramadol; Discogenic pain; Lumbar Discectomy
MeSH Terms: conditions — Intervertebral Disc Displacement | interventions — Tramadol; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tramadol (Active Comparator): Group Tramadol patients received tramadol 1 mg kg-1 iv
  Interventions: Drug: Tramadol
- Tramadol-Paracetamol (Active Comparator): Group Tramadol-Paracetamol patients received paracetamol 1 gr iv in addition to tramadol 1 mg kg-1 iv 30 minutes before the end of the operation and after the operation at 6 hour intervals for 24 hours
  Interventions: Drug: Tramadol; Drug: Paracetamol

INTERVENTIONS:
Drug: Tramadol — Tramadol iv
Drug: Paracetamol — Paracetamol iv
  Arms: Tramadol-Paracetamol

SUMMARY:
This study focused on to determine postoperative analgesic efficacy of tramadol compared to tramadol with addition of paracetamol after a lumbar disc surgery.

DETAILED DESCRIPTION:
Background:

Despite developments in treatment of pain, the availability of new drugs or increased knowledge of pain management, postoperative pain control after different surgeries still remains inadequate.

Aims:

This study focused on to determine postoperative analgesic efficacy of tramadol compared to tramadol with addition of paracetamol after a lumbar disc surgery.

Study Design:

In this study we have randomized 60 patients into two treatment groups. In Group Tramadol patients received tramadol, In Group TramadolParacetamol patients received paracetamol 1 gr iv in addition to tramadol 30 minutes before the operation ends and 1 g at 6 hour intervals.

Methods:

Severity of the pain, total tramadol consumption, adverse effects, ramsay sedation scale score, nausea/vomiting scores, patient satisfaction score were recorded in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

American Society of Anesthesiologists (ASA) 1 or 2 status patients with single level lumbar disc herniation.

Exclusion Criteria:

Patients who could not use a patient controlled analgesia (PCA) device, known allergies to any of the drugs used in this study,hepatic and renal dysfunction, herniated disc with neurological deficit or intense pain justifying emergency surgery and the patients whose body mass index is ≥30 kg/m2 were excluded from the study.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03-20 (Actual); Primary Completion 2015-01-12 (Actual); Study Completion 2015-04-03 (Actual)

PRIMARY OUTCOMES:
Severity of pain | 2 hours
  Self reported pain intensity

SECONDARY OUTCOMES:
Tramadol consumption | 2 hours
  Total tramadol consumption during time frame

CONTACTS AND LOCATIONS:
Overall Officials: Neslihan Uztüre, MD, Principal Investigator — Yeditepe University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Beakley BD, Kaye AM, Kaye AD. Tramadol, Pharmacology, Side Effects, and Serotonin Syndrome: A Review. Pain Physician. 2015 Jul-Aug;18(4):395-400. PMID 26218943
- [Background] Cakan T, Inan N, Culhaoglu S, Bakkal K, Basar H. Intravenous paracetamol improves the quality of postoperative analgesia but does not decrease narcotic requirements. J Neurosurg Anesthesiol. 2008 Jul;20(3):169-73. doi: 10.1097/ANA.0b013e3181705cfb. PMID 18580346
- [Background] Grundmann U, Wornle C, Biedler A, Kreuer S, Wrobel M, Wilhelm W. The efficacy of the non-opioid analgesics parecoxib, paracetamol and metamizol for postoperative pain relief after lumbar microdiscectomy. Anesth Analg. 2006 Jul;103(1):217-22, table of contents. doi: 10.1213/01.ane.0000221438.08990.06. PMID 16790656
- [Background] Hernandez-Palazon J, Tortosa JA, Martinez-Lage JF, Perez-Flores D. Intravenous administration of propacetamol reduces morphine consumption after spinal fusion surgery. Anesth Analg. 2001 Jun;92(6):1473-6. doi: 10.1097/00000539-200106000-00024. PMID 11375828
- [Background] Jirarattanaphochai K, Jung S. Nonsteroidal antiinflammatory drugs for postoperative pain management after lumbar spine surgery: a meta-analysis of randomized controlled trials. J Neurosurg Spine. 2008 Jul;9(1):22-31. doi: 10.3171/SPI/2008/9/7/022. PMID 18590407
- [Background] Kehlet H, Dahl JB. Anaesthesia, surgery, and challenges in postoperative recovery. Lancet. 2003 Dec 6;362(9399):1921-8. doi: 10.1016/S0140-6736(03)14966-5. PMID 14667752
- [Background] Korkmaz Dilmen O, Tunali Y, Cakmakkaya OS, Yentur E, Tutuncu AC, Tureci E, Bahar M. Efficacy of intravenous paracetamol, metamizol and lornoxicam on postoperative pain and morphine consumption after lumbar disc surgery. Eur J Anaesthesiol. 2010 May;27(5):428-32. doi: 10.1097/EJA.0b013e32833731a4. PMID 20173643
- [Background] Ohnesorge H, Bein B, Hanss R, Francksen H, Mayer L, Scholz J, Tonner PH. Paracetamol versus metamizol in the treatment of postoperative pain after breast surgery: a randomized, controlled trial. Eur J Anaesthesiol. 2009 Aug;26(8):648-53. doi: 10.1097/EJA.0b013e328329b0fd. PMID 19487950
- [Background] Olonisakin RP, Amanor-Boadu SD, Akinyemi AO. Morphine-sparing effect of intravenous paracetamol for post operative pain management following gynaecological surgery. Afr J Med Med Sci. 2012 Dec;41(4):429-36. PMID 23672109
- [Background] Pickering G, Loriot MA, Libert F, Eschalier A, Beaune P, Dubray C. Analgesic effect of acetaminophen in humans: first evidence of a central serotonergic mechanism. Clin Pharmacol Ther. 2006 Apr;79(4):371-8. doi: 10.1016/j.clpt.2005.12.307. PMID 16580905
- [Background] Remy C, Marret E, Bonnet F. Effects of acetaminophen on morphine side-effects and consumption after major surgery: meta-analysis of randomized controlled trials. Br J Anaesth. 2005 Apr;94(4):505-13. doi: 10.1093/bja/aei085. Epub 2005 Jan 28. PMID 15681586
- [Background] Shimia M, Parish M, Abedini N. The effect of intravenous paracetamol on postoperative pain after lumbar discectomy. Asian Spine J. 2014 Aug;8(4):400-4. doi: 10.4184/asj.2014.8.4.400. Epub 2014 Aug 19. PMID 25187855
- [Background] Sinatra RS, Jahr JS, Reynolds LW, Viscusi ER, Groudine SB, Payen-Champenois C. Efficacy and safety of single and repeated administration of 1 gram intravenous acetaminophen injection (paracetamol) for pain management after major orthopedic surgery. Anesthesiology. 2005 Apr;102(4):822-31. doi: 10.1097/00000542-200504000-00019. PMID 15791113
- [Background] Uzun S, Aycan IO, Erden IA, Sahin A, Aypar U. The addition of metamizole to morphine and paracetamol improves early postoperative analgesia and patient satisfaction after lumbar disc surgery. Turk Neurosurg. 2010 Jul;20(3):341-7. doi: 10.5137/1019-5149.JTN.3081-10.3. PMID 20669107
- [Background] Walder B, Schafer M, Henzi I, Tramer MR. Efficacy and safety of patient-controlled opioid analgesia for acute postoperative pain. A quantitative systematic review. Acta Anaesthesiol Scand. 2001 Aug;45(7):795-804. doi: 10.1034/j.1399-6576.2001.045007795.x. PMID 11472277
- [Background] White PF. Multimodal analgesia: its role in preventing postoperative pain. Curr Opin Investig Drugs. 2008 Jan;9(1):76-82. PMID 18183534
- [Background] White PF. The changing role of non-opioid analgesic techniques in the management of postoperative pain. Anesth Analg. 2005 Nov;101(5 Suppl):S5-S22. doi: 10.1213/01.ANE.0000177099.28914.A7. PMID 16334489
- [Background] Zhang Q, Qian J, Zhu Y. Meta-Analysis on Microdiscectomy and Sequestrectomy for Lumbar Disc Herniation. J Invest Surg. 2015;28(4):225-9. doi: 10.3109/08941939.2015.1006378. PMID 26268422